CLINICAL TRIAL: NCT06414161
Title: Management of Radiotherapy-related Xerostomia With Green Tea and Peppermint Oral Rinse: a Double-blind, Randomized Clinical Trial
Brief Title: Management of Radiotherapy-related Xerostomia With Green Tea and Peppermint
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: green tea and peppermint
Record Dates: First submitted 2024-04-19; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Radiation-induced Xerostomia
Keywords: xerostomia; green tea; pepprmint; Mucositis
MeSH Terms: conditions — Xerostomia; Mucositis | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: (Experimental): patients in test group will topically apply 20 ml (green tea plus peppermint) (1:1) to the oral mucosa. They will be instructed to keep green tea plus peppermint for at least 5 min duration and then to spit it out. They will be advised to rinse 20 mL of green tea plus peppermint in the same manner before sleeping from fourth week of radiotherapy to three months after radiotherapy.
  Interventions: Dietary Supplement: mix of (green tea and peppermint)
- Control group (Placebo Comparator): Patients in the control arm will topically apply 20 mL of 0.9% of saline 15 min before and after radiotherapy. They will be advised to rinse saline. They will be instructed to keep saline for at least 5 min duration and then to spit it out. They will be advised to rinse 20 mL of saline in the same manner before sleeping from fourth week of radiotherapy to three months after radiotherapy.
  Interventions: Dietary Supplement: mix of (green tea and peppermint)

INTERVENTIONS:
Dietary Supplement: mix of (green tea and peppermint) — Dried green tea leaves (100 gm) will be soaked into 500 ml of methanol solution for two days. The solution obtained will then be strained by a strainer and shifted to a glass plate. The plates will be left at room temperature from three to four days. Scraping out of the crystal powder of the extract from the plates will be carried out [27].
  The peppermint mouth rinse that was used in this study had 1% peppermint base, 10% xylisorb, 5% glycerin, 1% Tween 20%, 5% alcohol 96%, 0/18% methyl paraben, and 0/02% propyl paraben [28].
  Similarly, green tea plus peppermint mouthwash will be prepared at the same way but by adding 50% green tea leaves and 50% peppermint in the extract.

SUMMARY:
The goal of this study is to evaluate the clinical effectiveness of a mix of (green tea and peppermint) mouth rinse using the subjective dry mouth score as a primary objective and to assess the effect of that mix on the salivary flow rate and objective dry mouth score as a secondary objective.

DETAILED DESCRIPTION:
The Global Cancer Observatory from the World Health Organization estimates that head and neck cancer (HNC) incidence will reach approximately 1.5 million cases worldwide in 2020. Nevertheless, radiotherapy (RT) remains one of the cornerstone standard therapies to attenuate HNC progression. The advancement of linear accelerator (LINAC) technologies together with intensity-modulated radiation therapy (IMRT) techniques have enhanced the precision and efficiency of fractionated RT for HNC. Emerging research efforts have also been undertaken to understand these RT technologies' ability to spare the function of neighboring healthy tissues or organs like the salivary glands (SG).

Despite these research advances, a large majority of HNC patients who undergo RT display irreversible dry mouth symptoms (xerostomia) due to high radiation sensitivity of salivary gland (SG) secretory cells. This gland damage is thought to be triggered by an RT-induced loss of acinar cells and a potential impairment of the parasympathetic innervation and vascularization. Hence, the remaining integral SG stem/progenitor cells post-RT will define the true regenerative ability of the SG organ.

Cytoprotectant agents like amifostine have been recommended to prevent RT damage to SG cells. Amifostine is the only US Food and Drug Administration (FDA) approved drug for this prevention strategy. In Phase III clinical trials, amifostine was found to reduce xerostomia severity in subjects with grade two and above; however, more than 50% of subjects still presented acute xerostomia symptoms and oral mucosa inflammation. Moreover, amifostine has a very narrow therapeutic window. Therefore, frequent administration is required leading to severe side effects in more than half of the treated individuals. These side effects can lead to the discontinuation of amifostine treatment and RT delay in 25% of HNC patients. The high frequency of reported side effects and its high cost and low-quality evidence of efficacy from several clinical trials make amifostine a less promising pharmacological approach. Thus, novel pharmaceuticals are necessary to prevent SG damage and maintain the acinar epithelial and stem/progenitor cell populations in the SG organ.

In vitro and in vivo studies indicate green tea polyphenols (GTPs)/(-)-epigallocatechin-3-gallate (EGCG) as potential natural agents for xerostomia management, potentially delaying salivary dysfunction through molecular mechanisms. Researchers highlighted EGCG's role in suppressing autoantigens, influencing epithelial cell proliferation, and modulating antioxidant enzyme expression in salivary glands.

Peppermint essential oil is another herbal preparation with strong antibacterial and cooling effects. As a safe herbal preparation, peppermint essential oil has been found to be effective in alleviating the pain associated with aphthous stomatitis and managing dental plaque.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, aged above 20 years.
* All patients must have complaint of xerostomia.
* Objective dry mouth score from ( 2-5).
* Subjective dry mouth score from (1-4).
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Patient with history of any serious illness as malignancy.
* Patients with any autoimmune disease.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Subjective symptoms of oral dryness | Three points: -"baseline which is at the fourth week of radiotherapy", -"the second point is at seventh week of the radiotherapy, while the end point is after three months of radiotherapy.
  Using a questionnaire will be recorded according to the following:
  Q1. Does your mouth feel dry? Q2. Do you sip liquids to aid in swallowing dry food? Q3. Does your mouth feel dry when eating a meal? Q4. Does the amount of saliva in your mouth seem to be too little? Subject who answered affirmatively to at least one of the questions related to oral dryness will be considered as positive for subjective complaints of oral dryness.
  the score range frpm 1-4 according to the number of questions answered by yes

SECONDARY OUTCOMES:
Objective dry mouth score | Three points: -"baseline which is at the fourth week of radiotherapy", -"the second point is at seventh week of the radiotherapy, while the end point is after three months of radiotherapy.
  • The patients will be examined for their signs of dry mouth including: (Osailan et al., 2011).
  1. loss of pooled saliva
  2. Mouth mirror stickiness
  3. Stringy or foamy appearance
  4. Labial dehydration
  5. Irresponsiveness to parotid stimulation • Objective dry mouth scores will be calculated as the number of observed dry mouth signs (0-5), and patients with a score less than 2 will be excluded.

CONTACTS AND LOCATIONS:
Overall Officials: dalia Ghalwash, Study Director — professor
Locations (2):
- Egypt (2):
  - Ahmed Maher Teaching Hosipital, Cairo
  - ain shams University, Cairo

IPD SHARING:
Plan to Share IPD: No